CLINICAL TRIAL: NCT06986902
Title: Comparative Study Between the Effect of Nissen Fundoplication and Toupet Fundoplication on Post Operative Manometry Findings A Randomized Control Trial Study
Brief Title: Comparative Analysis of Postoperative Manometry Outcomes in Nissen vs Toupet Fundoplication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. IRB00006379
Record Dates: First submitted 2025-04-06; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-03

CONDITIONS: GERD - Gastro-Esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N GROUP (Experimental): Patients undergoing laparoscopic Nissen fundoplication (LNF), which involves a 360° total wrap of the gastric fundus around the esophagus.
  Interventions: Procedure: Laparoscopic Nissen Fundoplication
- T group (Experimental): Patients undergoing laparoscopic Toupet fundoplication (LTF), which involves a 270° posterior partial wrap of the gastric fundus around the esophagus.
  Interventions: Procedure: Laparoscopic Toupet fundoplication

INTERVENTIONS:
Procedure: Laparoscopic Nissen Fundoplication — a 360° total wrap of the gastric fundus around the esophagus.
  Arms: N GROUP
Procedure: Laparoscopic Toupet fundoplication — a 270° posterior partial wrap of the gastric fundus around the esophagus.
  Arms: T group

SUMMARY:
This randomized controlled trial investigates the effects of laparoscopic Nissen and Toupet fundoplication on postoperative esophageal manometry findings in patients with gastroesophageal reflux disease (GERD). The study, conducted at Ain Shams University Hospitals, involved 20 adult patients randomly assigned to undergo either procedure. Preoperative and postoperative high-resolution manometry (HRM) was used to assess lower esophageal sphincter (LES) pressure and esophageal motility.

DETAILED DESCRIPTION:
Preoperative Setting:

Before surgery, all patients underwent a thorough clinical assessment to evaluate the severity of their GERD symptoms, history of medication use, and the presence of extra-esophageal manifestations such as chronic cough or aspiration. A comprehensive diagnostic workup was conducted, including upper gastrointestinal endoscopy to assess mucosal integrity, rule out Barrett's esophagus, and evaluate the presence of a hiatal hernia. A barium swallow study was performed to assess esophageal motility, reflux severity, and anatomical abnormalities. The cornerstone of preoperative evaluation was high-resolution manometry (HRM), which provided precise measurements of lower esophageal sphincter (LES) pressure, esophageal peristalsis, and overall esophagogastric junction function.

Patients were deemed eligible for the study if they were between 18 and 65 years old and had documented low LES pressure on HRM. Those with persistent GERD symptoms despite at least 12 weeks of maximal medical therapy, intolerance to medication, or a desire to avoid lifelong proton pump inhibitor (PPI) therapy were considered suitable candidates. To ensure adequate postoperative esophageal motility, only patients with at least 30% esophageal peristalsis were included. Patients with esophageal motility disorders (such as achalasia), morbid obesity (BMI >35 kg/m²), a history of upper abdominal surgery, or a severely shortened esophagus were excluded. Patients classified as ASA III, IV, or V were also excluded due to the increased surgical risks associated with poor general health.

Patients were required to fast for at least 6-8 hours before surgery to minimize aspiration risk. Routine preoperative laboratory investigations, including a complete blood count (CBC), coagulation profile, and liver and kidney function tests, were performed. All patients underwent a pre-anesthesia assessment to determine their fitness for general anesthesia. On the day of surgery, prophylactic intravenous antibiotics were administered.

Intraoperative Setting:

The surgery was performed laparoscopically under general anesthesia. Patients were positioned in the modified lithotomy position with a reverse Trendelenburg tilt (head-up) to improve surgical exposure of the esophagogastric junction. The abdominal area was sterilized using antiseptic solution, and a CO₂ pneumoperitoneum was established (typically 12-15 mmHg) to facilitate laparoscopic access. A total of five to six laparoscopic ports were placed, with a 10-mm umbilical port for the camera and 5-mm ports for instruments and liver retraction.

For Nissen fundoplication, the procedure included circumferential dissection of the esophagus (ensuring 2-3 cm intra-abdominal length), crural closure with non-absorbable sutures, and mobilization of the gastric fundus (with division of short gastric vessels as needed). A 360° wrap was constructed and secured with four to five interrupted sutures. A 60F esophageal bougie was introduced intraoperatively to prevent a tight wrap.

For Toupet fundoplication, esophageal mobilization and crural closure were performed similarly. A 270° posterior wrap was constructed by positioning the gastric fundus posteriorly around the esophagus. It was secured with two to three sutures anchoring it to the right crura, two to three sutures attaching it to the esophagus, and two sutures securing it to the left crura. No esophageal bougie was used.

After the wrap, the surgeon ensured adequate tension, confirmed hemostasis, inspected for injury, and closed the abdominal incisions. Patients were extubated once fully recovered from anesthesia.

Postoperative Setting:

Following surgery, patients were monitored in the post-anesthesia care unit (PACU). Pain was managed with intravenous analgesics (e.g., paracetamol, NSAIDs, or opioids). Antiemetics such as ondansetron or metoclopramide were administered. Early ambulation was encouraged to reduce risks of deep vein thrombosis (DVT) and pulmonary complications.

Postoperative dietary advancement was structured to support healing. On the first postoperative day, patients were started on clear liquids. Over the next week, they progressed to a full liquid diet, then to soft/puréed foods by weeks 2-4, and finally to solids after four weeks while avoiding carbonated or hard foods.

All patients underwent high-resolution manometry (HRM) at six weeks postoperatively to assess LES pressure and esophageal motility. Data were collected and prepared for later analysis in accordance with study protocols.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 65 years of age
* Patients with pre-operable low LES pressure proven by High resolution manometry.
* Patients refractory to medical therapy: Persistent symptoms after 12 weeks of maximal medical therapies, recurrence upon cessation of medications.
* Patients who are non-compliance with medical therapies or inability to tolerate medical therapies .
* Patients with esophageal motility more than 30%

Exclusion Criteria:

* Patients with esophageal motility less than 30%.
* Patent with morbidly obese (BMI more than 35 kg/m2),
* Patients with recent upper abdominal surgery or severely shortened esophagus
* Extremes of age less than 18 and more than 65.
* Patients who are unfit for general anesthesia (ASAIII,IV or V)..

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Lower Esophageal Sphincter (LES) Resting Pressure | 6 Weeks Postoperative
  LES resting pressure will be recorded using high-resolution manometry (HRM) at 6 weeks after surgery to quantify baseline LES tone restoration.
  Unit of Measurment : mm Hg

OTHER OUTCOMES:
Distal Contractile Integral (DCI) | 6 Weeks Postoperative
  Postoperative peristaltic vigor will be quantified as DCI on HRM at 6 weeks. Unit of measurement : mm Hg·s·cm
Integrated Relaxation Pressure over 4 seconds (IRP-4s) | 6 Weeks Postoperative
  IRP-4s will be measured on HRM tracings 6 weeks postoperatively to assess adequacy of LES relaxation during swallowing.
  Unit of Measurment : mm Hg
Distal Latency | 6 Weeks Postoperative
  Time from swallow onset to distal contractile deceleration point will be recorded on HRM 6 weeks post-surgery.
  Unit of Measurment : seconds
Percentage of Normal Esophageal Contractions | 6 Weeks Postoperative
  Proportion of swallows exhibiting normal peristaltic patterns on HRM 6 weeks after surgery.
  unit of measurement : %
Percentage of Fragmented Esophageal Contractions | 6 Weeks Postoperative
  Proportion of swallows showing fragmented peristalsis on HRM 6 weeks post-operation.
  unit of measurement : %

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Gadalla, MS, Principal Investigator — Assistant lecturer in General surgery Department , Ain shams University Hospitals
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF